CLINICAL TRIAL: NCT06379308
Title: Anterior Cruciate Ligament (ACL) Revision Surgery: French National Study
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN552024/CHUSTE.
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: Knee; ACL; revision; surgery
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with Anterior Cruciate Ligament (ACL) revision: Patient with Anterior Cruciate Ligament (ACL) revision will be included. Questionary will be administrated and datas will be collected by medical record.
  Interventions: Other: questionaries; Other: datas of medical record

INTERVENTIONS:
Other: questionaries — Questionaries will be administered :
  * Anterior Cruciate Ligament Return to Sport and Injury (ACL-RSI)
  * Tegner Activity Scale (TAS)
  * Simple Knee Value (SKV)
  * International Knee Documentation Commitee (IKDC)
Other: datas of medical record — datas of medical record will be collected : epidemiological data, morphological data, operative data, clinical and functional outcomes, and surgical complication.

SUMMARY:
This is a national multicentric study led by the French Arthroscopy Society (SFA) evaluating clinical practice in anterior cruciate ligament (ACL) revision surgery (epidemiological data, morphological data, operative data, clinical and functional outcomes, and surgical complication rates).

ELIGIBILITY:
Inclusion Criteria:

* Patient with an anterior cruciate ligament (ACL) revision, defined as "all surgical procedures involving replacement of the anterior cruciate ligament (ACL) graft with a new graft".

Exclusion Criteria:

* multil-igament injuries
* any procedure where the ACL was not revised and where any additional graft was inserted
* Patients who had already undergone their first revision anterior cruciate ligament (ACL) procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with an anterior cruciate ligament (ACL) revision will be included.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Results of Functional score questionary Anterior Cruciate Ligament Return to Sport and Injury (ACL-RSI) | Months: 0, 6, 12 and 24
  Results of Functional score questionary Anterior Cruciate Ligament Return to Sport and Injury (ACL-RSI) will be analyzed.
  questionary Anterior Cruciate Ligament Return to Sport and Injury (ACL-RSI) has 12 questions (min = 0, max = 100). Greater psychological preparation is indicated by higher scores.
Results of Functional score questionary Tegner Activity Scale (TAS) | Months: 0, 6, 12 and 24
  Results of Functional score questionary Tegner Activity Scale (TAS) will be analyzed.
  The Tegner Activity Scale (TAS) is a scale of sporting and professional physical activities: from 0 (professional disability due to knee) to 10 (competitive sport such as soccer or rugby at national or international level).
Results of Functional score questionary Simple Knee Value (SKV) | Months: 0, 6, 12 and 24
  Results of Functional score questionary Simple Knee Value (SKV) will be analyzed.
  Scale from 0 to 100 to evaluate the knee function in daily life (0 is no function and 100 is normal function)
Results of Functional score questionary International Knee Documentation Commitee (IKDC) | Months: 0, 6, 12 and 24
  Results of Functional score questionary Knee Documentation Commitee (IKDC) will be analyzed.
  Subjective evaluation of the knee function (from 0 to 100%, 0 is no function and 100 is normal function)

SECONDARY OUTCOMES:
Surgical complications | From surgery to 2 months
  Report of surgical complications during the 2 months following the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Thomas NERI, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No